CLINICAL TRIAL: NCT03595579
Title: A Randomized, Double-Blind, Active-Controlled Trial of AXS-05 Administered Orally to Subjects With Major Depressive Disorder
Brief Title: Assessing Symptomatic Clinical Episodes in Depression
Acronym: ASCEND
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Axsome Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AXS-05-MDD-201
Record Dates: First submitted 2018-06-20; First posted 2018-07-23 (Actual); Results first posted 2021-09-24 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Major Depressive Disorder
Keywords: AXS-05; Major Depressive Disorder; MDD; Axsome; Depression; Dextromethorphan; Bupropion; Sigma-1; NDMA; ASCEND
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Bupropion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AXS-05 (Experimental)
  Interventions: Drug: AXS-05
- Bupropion (Active Comparator)
  Interventions: Drug: Bupropion

INTERVENTIONS:
Drug: AXS-05 — AXS-05 taken twice daily for 6 weeks.
  Arms: AXS-05
Drug: Bupropion — Bupropion taken twice daily for 6 weeks.
  Arms: Bupropion

SUMMARY:
Randomized, Double-Blind, Active-Controlled Study of AXS-05 for MDD.

DETAILED DESCRIPTION:
This study will evaluate the safety and efficacy of AXS-05 in a randomized, double-blind, active-controlled study in patients diagnosed with major depressive disorder (MDD) experiencing an acute episode.

ELIGIBILITY:
Inclusion Criteria:

* Currently meets DSM-5 criteria for MDD
* Body mass index (BMI) between 18 and 40 kg/m^2, inclusive
* Agree to use adequate method of contraception for the duration of the study
* Additional criteria may apply

Exclusion Criteria:

* Suicide risk
* History of treatment resistance in current depressive episode
* History of electroconvulsive therapy, vagus nerve stimulation, transcranial magnetic stimulation or any experimental central nervous system treatment during the current episode or in the past 6 months
* Pregnant, breastfeeding, or planning to become pregnant or breastfeed during the study
* Additional criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2018-05-30 (Actual); Primary Completion 2019-01-07 (Actual); Study Completion 2019-01-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Clinical Research Site, Beverly Hills, California
  - Clinical Research Site, Jacksonville, Florida
  - Clinical Research Site, Orlando, Florida
  - Clinical Research Site, Bellevue, Washington

IPD SHARING:
Plan to Share IPD: Yes
via publication

REFERENCES:
- [Derived] Tabuteau H, Jones A, Anderson A, Jacobson M, Iosifescu DV. Effect of AXS-05 (Dextromethorphan-Bupropion) in Major Depressive Disorder: A Randomized Double-Blind Controlled Trial. Am J Psychiatry. 2022 Jul;179(7):490-499. doi: 10.1176/appi.ajp.21080800. Epub 2022 May 18. PMID 35582785
- See also: Related Info — http://www.axsome.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AXS-05 | Bupropion
Started | 48 | 49
mITT Population | 43 | 37
Safety Population | 48 | 48
Completed | 38 | 35
Not Completed | 10 | 14

BASELINE CHARACTERISTICS:
Population: Participants randomized
Groups:
- Total: Total of all reporting groups
Arm/Group | AXS-05 | Bupropion | Total
Number analyzed (Participants) | 48 | 49 | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.8 (11.98) | 39.9 (12.96) | 39.1 (12.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 32 | 60
  Male | 20 | 17 | 37
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 16 | 31
  White | 32 | 29 | 61
  More than one race | 0 | 4 | 4
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: MADRS Score - Overall Change From Baseline
Description: The primary objective of the study was to assess the effect of AXS-05 versus bupropion as measured by the Montgomery-Åsberg Depression Rating Scale (MADRS) for change in severity of depressive symptoms. The MADRS is a 10-item scale and items are scored between 0-6 points. For each item, a score of 0 indicates the absence of symptoms, and a score of 6 indicates symptoms of maximum severity. A maximum total score is 60 points.
Time Frame: Assessed at week 1, 2, 3, 4, 5 and 6 (averaged over the entire 6-week treatment period)
Population: modified Intent-to-Treat (mITT) Population
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | AXS-05 | Bupropion
Number analyzed (Participants) | 43 | 37
score on a scale | 13.7 (0.63) | 8.8 (0.68)
Statistical Analysis 1: Comparison: AXS-05 vs Bupropion; Test type: Superiority; p < .001, Mixed Models Analysis

2. Other Pre Specified Outcome: MADRS Score - Change From Baseline to Week 6
Description: as for outcome 1
Time Frame: 6 weeks
Population: modified Intent-to-Treat (mITT) Population
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | AXS-05 | Bupropion
Number analyzed (Participants) | 43 | 37
score on a scale | 17.2 (1.4) | 12.1 (1.5)
Statistical Analysis 1: Comparison: AXS-05 vs Bupropion; Test type: Superiority; p = 0.013, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of signing the ICF through 30 days after the last study visit or Early Termination (ET), whichever occurred first, an average of 11 weeks per participant.
Description: Safety Population
Arm/Group | AXS-05 | Bupropion
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/48
Other Adverse Events (participants affected / at risk) | 35/48 | 30/48
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AXS-05 (N=48) | Bupropion (N=48)
Constipation (Gastrointestinal disorders) | 3 | 4
Diarrhea (Gastrointestinal disorders) | 3 | 4
Dry mouth (Gastrointestinal disorders) | 5 | 4
Nausea (Gastrointestinal disorders) | 8 | 6
Decreased appetite (Metabolism and nutrition disorders) | 5 | 4
Dizziness (Nervous system disorders) | 10 | 2
Headache (Nervous system disorders) | 4 | 5
Sedation (Nervous system disorders) | 3 | 0
Tension headache (Nervous system disorders) | 3 | 2
Anxiety (Psychiatric disorders) | 5 | 1
Insomnia (Psychiatric disorders) | 4 | 2
Yawning (Respiratory, thoracic and mediastinal disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-06-28): https://cdn.clinicaltrials.gov/large-docs/79/NCT03595579/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-11): https://cdn.clinicaltrials.gov/large-docs/79/NCT03595579/SAP_001.pdf